CLINICAL TRIAL: NCT06671340
Title: Effects of Repeated Dose of Dorzagliatin on Insulin Secretion, Glucagon Release and Incretin Function in Intermediate Hyperglycemia and Type 2 Diabetes
Brief Title: Chronic Dorzagliatin on Insulin and Incretin Function in Intermediate Hyperglycemia and Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elaine Chow (Other)
Responsible Party: Sponsor-Investigator, Elaine Chow, Clinical Associate Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENSITISE-3
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus; Prediabetes / Type 2 Diabetes
Keywords: clamp; diabetes; glucokinase activator
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IH/T2D (Experimental): partipiants with intermediate hyperglycemia (IH) n=15 or T2D (n=15)
  Interventions: Drug: Dorzagliatin

INTERVENTIONS:
Drug: Dorzagliatin — chronic treatment with dorzagliatin for 4 weeks (50mg twice daily or 75mg twice daily, oral)

SUMMARY:
A total of 30 subjects will be recruited 15 with intermediate hyperglycemia and 15 in the tyep 2 diabetes group respectively. Eligible participants will undergo hyperglycemic-clamp/oral glucose tolerance at baseline and after 4 weeks of dorzagliatin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged ≥ 18 years but < 70 years
2. Male or female
3. Body mass index of over 18 kg/m2 and < 35 kg/m2

Additional inclusion criteria for IH group

* Fasting plasma glucose <7.0 mmol/L and HbA1c < 6.5%
* 1 hour plasma glucose ≥8.6 and <11.6 mmol/L on 75g oral glucose tolerance test (OGTT)
* No use of glucose lowering drugs in past 6 months

Additional inclusion criteria for T2D group

* HbA1c 6.5 to 10% at screening
* On diet control, or stable dose of oral glucose lowering drugs metformin for at least 8 weeks

Exclusion Criteria:

* 1. Subjects who do not agree to participate in this study. 2. Country of birth is unknown. 3. Body weight less than 45kg. 4. Acute phase of cerebrovascular and cardiovascular diseases (within 6 months of recruitment).

  5. Subjects with severe renal dysfunction as defined by eGFR <30 ml/min/1.73m2 or patients receiving renal dialysis (such as haemodialysis or continuous ambulatory peritoneal dialysis).

  6. Severe hepatic dysfunction as defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times upper limit of normal.

  7. Severe cardiovascular disease, history of stroke, heart failure (NYHA III or IV) or history of myocardial infarction within last 12 months.

  8. History of drug abuse or excessive alcohol intake based on investigator judgment.

  9. Dehydration, diarrhoea or vomiting at the time of recruitment. 10. Subjects with severe infection, in perioperative period or with serious injury at the time of recruitment.

  11. Subjects with anaemia (Haemoglobin <9.0mg/dL). 12. Pregnant or lactating or intending to become pregnant within 30 days after last dose of study drug.

  13. Participation in a clinical trial with investigational product within 30 days before enrolment.

  14. Donation or loss of blood (excluding the volume of blood that will be drawn during screening procedures) as follows: ≥300 mL of blood within 30 days prior to study drug administration.

  15. Subjects judged unsuitable for the study based on investigator judgment. 16. Use of strong or moderate CYP3A4 inhibitors or inducers and cannot be discontinued.

  17. Unwilling or unable to follow protocol requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Acute Insulin secretion | At baseline and after 4 weeks of study drug treatment
  Acute (first phase) insulin response (AIRg) to glucose will be calculated as the mean incremental responses above baseline (average of -20 and -10 and 0 minutes) to the samples drawn at 2, 4, 6, 8 and 10 minutes of the hyperglycemic clamp.

SECONDARY OUTCOMES:
Second phase insulin secretion | At baseline and after 4 weeks of study drug treatment
  The mean incremental insulin levels between 60 to 90 minutes of hyperglycemic clamp
Beta cell glucose sensitivity | At baseline and after 4 weeks of study drug treatment
  Beta cell glucose sensitivity will be calculated as increment of insulin secretion in 60-90 minutes of the clamp minus basal insulin divided by glucose change in the same period
Glucagon-like peptide -1 (GLP-1) | At baseline and after 4 weeks of study drug treatment
  GLP-1 secretion Area under the curve (0-270 minute during hyperglyemic- OGTT clamp study)
Glucagon | At baseline and after 4 weeks of study drug treatment
  Glucagon area under the curve (0-270 minute) during hyperglyemic- OGTT clamp
Incretin effect | At baseline and after 4 weeks of study drug treatment
  Difference between the post prandial (100-270min) and preprandial (60-90min) C peptide response

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, MBChB, PhD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Phase 1 Clinical Trial Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes